CLINICAL TRIAL: NCT00179504
Title: The Effect of Relaxation Response Training on Declarative Memory and Learning in High School Students
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 2001-P-000110
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2007-11-05 (Estimated); Status verified 2007-11

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Outcomes Assessor

INTERVENTIONS:
Behavioral: Relaxation Response — Relaxation training

SUMMARY:
Stress contributes to health and behavioral issues in students, but will not be integrated into schools without evidence of benefit. This study was conducted to determine if a 6-week relaxation response (RR) curriculum improves cognitive performance in ninth grade students.

DETAILED DESCRIPTION:
Stress contributes to health and behavioral issues in students, but will not be integrated into schools without evidence of benefit. This study was conducted to determine if a 6-week relaxation response (RR) curriculum improves cognitive performance in ninth grade students.

ELIGIBILITY:
Inclusion Criteria:

* a member of 9th grade at a residential preparatory school.

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2000-07; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Determine if a 6-week relaxation response (RR) curriculum improves cognitive performance. | 6 weeks

SECONDARY OUTCOMES:
Evaluate whether the program would influence levels of salivary cortisol and whether there would be a correlation between cortisol levels and performance on the cognitive tasks. | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery A Dusek, PhD, Principal Investigator — Beth Israel Deaconess Medical Center, Mind/Body Medical Institute